CLINICAL TRIAL: NCT00569049
Title: Molecular Analysis of Breast Cancer
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of California (Other); California Breast Cancer Research Program (Other); Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: SU-11052007-799; 1028313-100-JAACC; 1045090-101-KBAHQ; 10EB-10086; 11IB-0175; CA085129; 1R01CA109325-01; 8EB-1106; BRSNSTU0001 (Other: Stanford OnCore)
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Breast Cancer Non-invasive Breast Cancer; Breast Cancer Early Stage Breast Cancer (Stage 1-3)
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tumor, normal tissue and blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: breast tissue, lymph node tissue or blood — Molecular Analyses of samples

SUMMARY:
This is a research-based study that is looking at the biologic features of breast tissue, lymph node tissue, or blood in order to study breast cancer development growth, and spread. Through tissue and/or blood samples we hope to gain further knowledge and understanding of how to improve diagnosis and treatment of breast cancer by identifying the molecular markers that predict clinical outcome and response to therapy.

DETAILED DESCRIPTION:
The tissue obtained in this protocol will be used for genome-wide examination of DNA, RNA expression profiling, proteomic analyses, isolation and analyses of normal and cancer stem cells, isolation and analyses of circulating tumor cells, possible analyses of immune cells, and possible analyses of serum factors. The tissue may also be used to develop patient-specific cell culture models or mouse xenograft models of breast cancer for biologic study of tumor progression and metastases and for therapeutic testing. In general, the tissue will be used in studies that will molecularly classify tumors, identify prognostic markers, identify potential therapeutic markers, identify potential treatment targets, and help us better understand the biology and specific role played by different tumor cells in the metastatic process.

The ultimate goal is to use molecular analyses to improve the diagnosis and treatment of breast cancer.

ELIGIBILITY:
Inclusion Criteria:People eligible for this study include anyone older than 18 years who is undergoing one of the following procedures: core needle or surgical breast biopsy, lumpectomy, mastectomy, axillary lymph node surgery, breast reduction surgery, or ductal lavage or ductoscopy. Patients who have had breast cancer in the past who are currently free of disease or who have a breast cancer recurrence are also eligible. All patients who participate must be able to understand and sign the informed consent. Although most patients will be female, any males undergoing the above procedures are also eligible for this study. Exclusion Criteria:Any patient who is less than 18 years old, who is unable to understand the informed consent, or not undergoing the above procedures will be excluded from this research.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients undergoing breast cancer procedures
Sampling Method: Non-Probability Sample
Enrollment: 788 (Actual)
Dates: Start 1996-05; Primary Completion 2011-07-01 (Actual); Study Completion 2011-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Curtis, PhD, MSc, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States